CLINICAL TRIAL: NCT07018674
Title: Evaluation of Acute Cognitive Effects of Brain Edge on Healthy Volunteers
Brief Title: Acute Cognitive Effects of Brain Edge
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nature's Sunshine Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NSP-CT-023
Record Dates: First submitted 2025-05-14; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Cognitive Health; Mood
MeSH Terms: interventions — Water

STUDY DESIGN:
Intervention Model Description: Double Blind Placebo Controlled
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crossover Arm 1: Brain Edge then Placebo (Experimental): Participants will receive Water during Visit 1, Brain Edge during Visit 2, and the Placebo on Visit 3
  Interventions: Dietary Supplement: Experimental; Other: Placebo; Other: Water
- Crossover Arm 2: Placebo then Brain Edge (Experimental): Participants will receive Water during visit 1, the Placebo during Visit 2, and Brain Edge during Visit 3
  Interventions: Dietary Supplement: Experimental; Other: Placebo; Other: Water

INTERVENTIONS:
Dietary Supplement: Experimental — Brain Edge, a cognition supporting supplement beverage formulated from herbs, vitamins, and amino acids.
Other: Placebo — A sensory-matched placebo beverage formulated from flavors, colors, fillers, and excipients.
Other: Water — Bottled Water

SUMMARY:
A double-blind placebo-controlled crossover study exploring the cognitive effects of Brain Edge; a supplement consisting of a blend of herbs and amino acids. 50 healthy adult subjects will be evaluated over 3 sessions. Evaluation of cognitive performance will be determined by computer-based software, surveys, and VR headset experiences.

DETAILED DESCRIPTION:
Clinical visits will take place in the mornings over 3 days. Subjects will meet with principal investigator or study staff at all clinical visits. During the clinical visits, the study clinician will assess for signs and symptoms of adverse events, dispense study products, administer the cognitive tests, and answer any questions from the subjects.

Visit 1 is characterized by subject screening, familiarizing participants with the cognitive tests, and establishing baseline performance values. After Subject Consent has been obtained, subjects will be assigned a Subject Identification Number (ID) and be randomly assigned to a study arm.

1. For subjects of childbearing potential, a urine pregnancy test (UPT) will be administered to ensure the subject is not pregnant.
2. Subjects will fill out the Entry Survey on a computer tablet.
3. Subjects will participate in the PEBL testing battery on a laptop using a keyboard and mouse. The battery includes the following tests:

   1. Matrix Pattern Rotation
   2. Stroop Task
   3. Sternberg Scanning Task
   4. Berg Wisconsin Card Sorting
   5. 9-Cell reaction test
   6. Math Test
4. Subject will be offered some water to drink. On visit 2 and 3, study staff will provide subject with a prepared sample of either Brain Edge, or Placebo. Samples will be administered in a double blinded manner.
5. Subjects will use the VR headset to play 3 songs in Beat Saber.

   1. Rum N Bass
   2. Burning Sands
   3. A song designated by study staff.
6. Subjects will fill out the Visit 1 Mid-Visit Snapshot Survey on a computer tablet.
7. Next, subjects will again participate in the PEBL testing battery using a mouse and keyboard. The tests will be the same as before.
8. The participant will again use the VR headset to play some songs. 2 of the songs will be the same as previous (Rum N Bass and Burning Sands), while the third song will be different.
9. Each participant will then be given the Visit Exit survey to fill out. Principal investigator or study staff will be available to provide explanations for the tests, answer any questions about the study or product, and to provide technical support for any of the devices. The test results from this day will provide a set of baseline values that will be used as a reference point for the tests on subsequent days.

Visit 2 marks the beginning of the experimental crossover portion of the study. Principal investigator or Study staff will answer questions and resolve subjects' concerns as needed.

Subjects will repeat the same testing procedures as the previous visit, with the addition of taking either the placebo or the Brain Edge sample immediately before playing the first round of Beat Saber. Samples will be double blinded.

Visit 3 will be the crossover portion of the study. If participants received a placebo during visit 2, the study sample for visit 3 will be Brain Edge. Conversely, those who received Brain Edge during visit 2 will receive a placebo during visit 3. Study testing procedures will proceed in the same manner as previous visits.

Visit 3 is the final visit of the study. However, to ensure that all adverse events are captured and recorded, subjects will be asked to fill out a final survey on the day following their last visit.

ELIGIBILITY:
Inclusion Criteria:

* Men, women and non-binary adults, ≥18 and <60 years old
* Generally healthy
* Ability to understand and the willingness to follow the study procedures.
* Willing to maintain a consistent diet (including medications, vitamins and supplements) and lifestyle routine throughout the study.
* Willing to give written informed consent to participate in the study.

Exclusion Criteria:

* Pregnant or nursing.
* Minors below the age of majority.
* Taking any prescription stimulants or anxiolytics.
* Typical caffeine intake above 250 mg/day.
* Neurological conditions including epilepsy, color blindness, ADD / ADHD, Learning disabilities, or dementia.
* Change in prescription, non-prescription, nutritional supplements and/or medical foods within 7 days prior to Day 1 and for the duration of the study.
* Use of prescriptions medications and/or nonprescription medications for acute and semi-acute medical conditions 30 days prior to Day 1 and for the duration of the study.
* Use of an investigational drug or participation in an investigational study within 30 days prior to Day 1 and for the duration of the study.
* Routine use of high dose caffeine >250mg products within 7 days prior to Day 1 and for the duration of the study.
* Subjects with a history of allergy or intolerance to any ingredient in study product. Specific details of each product will be included in the formal Study Informed Consent.
* Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, endocrinologic, neurologic, immunologic, or hematologic disease.
* Subjects with a current diagnosis or personal history of:
* Any cardiovascular disease including myocardial infarction, angina, cardiovascular surgery, congestive heart failure, cardiac arrhythmias or conduction abnormalities, cerebrovascular accident, transient ischemic attack (TIA), or peripheral vascular disease, deep vein thrombosis or pulmonary embolus.
* Any neurological condition including ADD, ADHD, Epilepsy, Narcolepsy, insomnia, or autism spectrum disorders.
* Any serious mental illness including a history of attempted suicide.
* Use of drugs of abuse (such as marijuana, cocaine, opiates and methamphetamine) 7 days prior to Day 1 and for the duration of the study.
* Inability to comply with study and/or follow-up visits.
* Any concurrent condition (including clinically significant abnormalities in medical history, physical examination, or laboratory evaluations) which, in the opinion of the PI, would preclude safe participation in this study or interfere with compliance.
* Any sound medical, psychiatric and/or social reason which, in the opinion of the PI, would preclude safe participation in this Study or interfere with compliance.

Co-enrollment in other trials is restricted other than for observational studies. Study staff should be notified of co-enrollment as it may require the approval of the investigator.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with supplementation-related adverse events (AEs) as assessed by Common Terminology Criteria for Adverse Events v4.0 (CTCAE v4.0). | 7 days after final clinical visit
  Data collected at individual study visits will be used to assess participants for any adverse events associated with the study procedures or products. Subjects with ongoing adverse events will be followed until resolution at the discretion of the PI.

SECONDARY OUTCOMES:
Attention Shifting | Prior to supplementation (Baseline) and 30 minutes after supplementation (Post) during each of the 3 clinical visits.
  Assessed by changes in attention shifting score in the Berg-Wisconsin Card Sorting Task Test.
Working Memory | Prior to supplementation (Baseline) and 30 minutes after supplementation (Post) during each of the 3 clinical visits.
  Assessed by changes in score in Sternberg Scanning Task Test.
Reaction Time | Prior to supplementation (Baseline) and 30 minutes after supplementation (Post) during each of the 3 clinical visits.
  Assessed by changes in score in 9-cell reaction test.
Selective Attention | Prior to supplementation (Baseline) and 30 minutes after supplementation (Post) during each of the 3 clinical visits.
  Assessed by changes in score in Stroop Task Test.
Executive Function | Prior to supplementation (Baseline) and 30 minutes after supplementation (Post) during each of the 3 clinical visits.
  Assessed by a change in scores in a simple mathematics test
Visual Processing | Prior to supplementation (Baseline) and 30 minutes after supplementation (Post) during each of the 3 clinical visits.
  Assessed by score in Matrix Rotation Test
Gaming Performance | Prior to supplementation (Baseline) and 60 minutes after supplementation (Post) during each of the 3 clinical visits.
  Assessed by score changes in Beat Saber (Virtual Reality Rhythm game).
Subjective Mood and Emotional State | Prior to Supplementation (Baseline), 30 minutes after supplementation (Midpoint) and approximately 90 minutes after supplementation (Post) on each of the 3 clinical visits.
  Assessed by relative changes in scored survey question results.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Lamb, MD, Principal Investigator — Nature's Sunshine Products, Inc.
Locations (1):
- The Hughes Center for Research and Innovation, Lehi, Utah, United States

IPD SHARING:
Plan to Share IPD: No